CLINICAL TRIAL: NCT03581097
Title: The Effect of Informational Videos on Preoperative Anxiety and Satisfaction Levels in Patients Undergoing Elective Ambulatory Surgery. A Case-control Clinical Trial
Brief Title: Educational Video and Peri-operative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Samuele Ceruti, Dr. med., University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CERU-1801
Record Dates: First submitted 2018-06-13; First posted 2018-07-10 (Actual); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Ambulatory Surgical Procedures; Anxiety Disorders
Keywords: Anxiety disorders; hand surgery; Educational Video
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Retrospective, single centre, case-control trial
Who Masked: Investigator
Masking Description: Surgeon and investigators involved in subsequent data analysis were blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Patients in the film group watched the film using a laptop computer equipped with headphones, and Visual Analog Pain Scale (VAS) was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of intravenous regional anesthesia
  Interventions: Other: Video Group
- Control Group (No Intervention): Patients assigned to this control group were not shown the video and underwent an otherwise identical preoperative preparation procedure.

INTERVENTIONS:
Other: Video Group — Patients in the film group watched the film using a laptop computer equipped with headphones, and Visual Analog Pain Scale (VAS) was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of Intra-Venous Regional Anesthesia (IVRA)
  Arms: Video Group

SUMMARY:
Preoperative anxiety is a common problem with an impact on surgical outcome, anaesthetic drug dosage and patient's satisfaction. An important component of preoperative anxiety is due to concerns related to anaesthesia. Appropriate patients information has been shown to reduce preoperative anxiety level and this can be effectively achieved through a video. The aim of this study is to assess the impact of an informative video about the anaesthesia technique on patient's preoperative anxiety levels before minor ambulatory procedures.

The study design is a prospective, randomized, controlled clinical trial, where we use of short patient educational video to reduce preoperative anxiety level, explaining all sequence of major events between the arrival in the operating room and the performance of anaesthesia.

DETAILED DESCRIPTION:
Anxiety is a common problem in patients undergoing invasive procedures, arriving in some studies up to 60-80%. Perioperative anxiety is correlated with hemodynamic effects (such as arterial hypertension and arrhythmias), it can have an impact on final surgical outcome, on anaesthetics drug dosage, and also with an growth about the perception of post-operative pain, leading to a substantial increase in analgesics dose and the number of post-operative hospitalization days. Finally, perioperative anxiety can reduce the patient's overall satisfaction with the quality of perioperative care.

Patients' satisfaction is largely based on their expectations and it forms part of the surgeon's reward: satisfied patients are more likely to maintain a good relationship with the surgeon, abstain from so called "doctor shopping", avoid malpractice litigations and recommend their surgeon to others. Last but not least, satisfied patients are more likely to comply with postoperative prescriptions and attend follow-up appointments. In non-life threatening procedures however, the main source of preoperative anxiety is often the outlook of anaesthesia rather than surgery itself, this being mainly related to a lack of enough information about the anaesthetic procedure. These fears are largely underestimated in routine minor procedures (such as ambulatory surgery) and thus risk to be not properly addressed. Due to lack of time and resources, this could have a significant impact on global patient satisfaction. Also if major complications (e.g. cardiac mortality) are surgery-related, anxiety is also associated with poor surgical outcome. How to identify and treat patients who will likely benefit from more information about anaesthesia is an important question that remains relatively unaddressed. However, it's known that more information about surgery reduces the level of anxiety and apprehension.

Some strategies have been developed to try to reduce pre-operative stress: deliver clinical information has proven to be able to relieve patient anxiety. Written information has recognised useful, but not all patients have shown the same degree of culture needed to read and understand texts. The use of multimedia information (such as videos) has already been studied and some trials have shown a certain anxiolytic effect, but data are conflicting. A part of this disparity probably derives from differences in methodology and culture between patients.

For these reasons the investigators developed a trial using a short educational video about the global management of local anaesthesia on outpatient hand surgery. The aim of this study is to assess the impact of this educational video about perioperative patient's anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years,
* American Society Anesthesiology (ASA) score I-III patients
* patients undergoing elective hand-surgery operation
* patients anesthetized by IntraVenous Regional Anesthesia (IVRA)

Exclusion Criteria:

* patient refusal,
* on-going anxiolytic or anti-depressive therapy,
* diagnosis of anxiety or psychiatric disorders,
* general contraindications to IVRA,
* limited compliance
* language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2018-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Fusetti, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Andrea Saporito MD, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Bandeira D, Ferreira MB. Risk factors for preoperative anxiety in adults. Acta Anaesthesiol Scand. 2001 Mar;45(3):298-307. doi: 10.1034/j.1399-6576.2001.045003298.x. PMID 11207465
- [Background] Edward GM, v d Naald N, Oort FJ, de Haes HC, Biervliet JD, Hollmann MW, Preckel B. Information gain in patients using a multimedia website with tailored information on anaesthesia. Br J Anaesth. 2011 Mar;106(3):319-24. doi: 10.1093/bja/aeq360. Epub 2010 Dec 10. PMID 21149288
- [Background] Grossi G, Perski A, Feleke E, Jakobson U. State anxiety predicts poor psychosocial outcome after coronary bypass surgery. Int J Behav Med. 1998;5(1):1-16. doi: 10.1207/s15327558ijbm0501_1. PMID 16250712
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Morgan J, Roufeil L, Kaushik S, Bassett M. Influence of coping style and precolonoscopy information on pain and anxiety of colonoscopy. Gastrointest Endosc. 1998 Aug;48(2):119-27. doi: 10.1016/s0016-5107(98)70152-x. PMID 9717776
- [Background] Ramsay MA. A survey of pre-operative fear. Anaesthesia. 1972 Oct;27(4):396-402. doi: 10.1111/j.1365-2044.1972.tb08244.x. No abstract available. PMID 4634747
- [Background] Sorlie T, Busund R, Sexton J, Sexton H, Sorlie D. Video information combined with individualized information sessions: Effects upon emotional well-being following coronary artery bypass surgery--A randomized trial. Patient Educ Couns. 2007 Feb;65(2):180-8. doi: 10.1016/j.pec.2006.07.006. Epub 2006 Sep 7. PMID 16959466
- [Background] Takahashi Y, Tanaka H, Kinjo M, Sakumoto K. Prospective evaluation of factors predicting difficulty and pain during sedation-free colonoscopy. Dis Colon Rectum. 2005 Jun;48(6):1295-300. doi: 10.1007/s10350-004-0940-1. PMID 15793639
- [Result] Arabul M, Kandemir A, Celik M, Alper E, Akpinar Z, Aslan F, Vatansever S, Unsal B. Impact of an information video before colonoscopy on patient satisfaction and anxiety. Turk J Gastroenterol. 2012;23(5):523-9. doi: 10.4318/tjg.2012.0416. PMID 23161296
- [Result] Ayral X, Gicquere C, Duhalde A, Boucheny D, Dougados M. Effects of video information on preoperative anxiety level and tolerability of joint lavage in knee osteoarthritis. Arthritis Rheum. 2002 Aug;47(4):380-2. doi: 10.1002/art.10559. PMID 12209483
- [Result] Badner NH, Nielson WR, Munk S, Kwiatkowska C, Gelb AW. Preoperative anxiety: detection and contributing factors. Can J Anaesth. 1990 May;37(4 Pt 1):444-7. doi: 10.1007/BF03005624. PMID 2340614
- [Result] Danino AM, Chahraoui K, Frachebois L, Jebrane A, Moutel G, Herve C, Malka G. Effects of an informational CD-ROM on anxiety and knowledge before aesthetic surgery: a randomised trial. Br J Plast Surg. 2005 Apr;58(3):379-83. doi: 10.1016/j.bjps.2004.10.020. PMID 15780234
- [Result] Cornoiu A, Beischer AD, Donnan L, Graves S, de Steiger R. Multimedia patient education to assist the informed consent process for knee arthroscopy. ANZ J Surg. 2011 Mar;81(3):176-80. doi: 10.1111/j.1445-2197.2010.05487.x. Epub 2010 Oct 1. PMID 21342392
- [Result] Crabtree TD, Puri V, Bell JM, Bontumasi N, Patterson GA, Kreisel D, Krupnick AS, Meyers BF. Outcomes and perception of lung surgery with implementation of a patient video education module: a prospective cohort study. J Am Coll Surg. 2012 May;214(5):816-21.e2. doi: 10.1016/j.jamcollsurg.2012.01.047. Epub 2012 Mar 28. PMID 22464659
- [Result] Eley VA, Searles T, Donovan K, Walters E. Effect of an anaesthesia information video on preoperative maternal anxiety and postoperative satisfaction in elective caesarean section: a prospective randomised trial. Anaesth Intensive Care. 2013 Nov;41(6):774-81. doi: 10.1177/0310057X1304100613. PMID 24180719
- [Result] Hering K, Harvan J, Dangelo M, Jasinski D. The use of a computer website prior to scheduled surgery (a pilot study): impact on patient information, acquisition, anxiety level, and overall satisfaction with anesthesia care. AANA J. 2005 Feb;73(1):29-33. PMID 15727280
- [Result] Herrmann KS, Kreuzer H. A randomized prospective study on anxiety reduction by preparatory disclosure with and without video film show about a planned heart catheterization. Eur Heart J. 1989 Aug;10(8):753-7. doi: 10.1093/oxfordjournals.eurheartj.a059560. PMID 2792117
- [Result] Jlala HA, French JL, Foxall GL, Hardman JG, Bedforth NM. Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia. Br J Anaesth. 2010 Mar;104(3):369-74. doi: 10.1093/bja/aeq002. Epub 2010 Feb 1. PMID 20124283
- [Result] Jones MP, Ebert CC, Sloan T, Spanier J, Bansal A, Howden CW, Vanagunas AD. Patient anxiety and elective gastrointestinal endoscopy. J Clin Gastroenterol. 2004 Jan;38(1):35-40. doi: 10.1097/00004836-200401000-00009. PMID 14679325
- [Result] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Result] Pager CK. Randomised controlled trial of preoperative information to improve satisfaction with cataract surgery. Br J Ophthalmol. 2005 Jan;89(1):10-3. doi: 10.1136/bjo.2004.048637. PMID 15615737
- [Result] Zieren J, Menenakos C, Mueller JM. Does an informative video before inguinal hernia surgical repair influence postoperative quality of life? Results of a prospective randomized study. Qual Life Res. 2007 Jun;16(5):725-9. doi: 10.1007/s11136-007-9171-y. Epub 2007 Feb 8. PMID 17286194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A consecutive cohort of adult patients scheduled for elective ambulatory hand surgery of less than one-hour duration with an intravenous regional anesthesia was recruited
Pre-assignment Details: Patients were randomized with a free web tool (available at www.randomizer.org) in a consecutive order into two parallels groups
Groups:
- Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and VAS score was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of intravenous regional anesthesia
  Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and VAS score was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the OR and the performance of IVRA
Period: Overall Study
Arm/Group | Video Group | Control Group
Started | 46 | 47
Completed | 46 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: During the 8 months long study period, a total of 152 consecutive patients met the inclusion criteria and were successfully enrolled in the study protocol. Of these, 59 patients were excluded due to the use of anxiolytics medications; 93 patients were then included into the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Group | Control Group | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.8) | 54.8 (14.4) | 55.65 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 19 | 24 | 43
Right-hand dominance [Count of Participants; unit: Participants] | 42 | 43 | 85
Systolic arterial pressure [Mean (Standard Deviation); unit: mmHg] | 139.4 (22.1) | 129.2 (17.8) | 134.3 (19.95)
Diastolic arterial pressure [Mean (Standard Deviation); unit: mmHg] | 81.7 (10.9) | 78.4 (10.1) | 80.05 (10.5)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 75.4 (13.1) | 71.8 (10.2) | 73.6 (11.65)
Breath rate [Mean (Standard Deviation); unit: Breath per minute] | 14.7 (3.1) | 13.8 (1.5) | 14.25 (2.3)
Basal anxiety level [Mean (Standard Deviation); unit: units on a scale] — The VAS score (Visual Analogue Scale) is an instrument used for measuring anxiety. It's a semi-quantitative visual scale (from 0 - no anxiety - to 5 - maximal anxiety) that is used to measure patients' anxiety levels, asking each patient to subjectively quantify its own anxiety.
  units on a scale | 1.2 (1.1) | 1.0 (1.2) | 1.1 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: VAS-A Score Anxiety Level (Adapted Visual-Analogue Scale)
Description: Primary outcome measure is to see and analyze any difference in preoperative anxiety between the video and control group, measured on our Adapted Visual Analogue Scale (VAS-A). Scale range is 0 to 5, where 0 means no anxiety, while 5 means maximal anxiety. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of regional anesthesia.
Time Frame: 2 hours
Population: Anxiety level measured on admission in the day-hospital clinic
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and Visual Analog Pain Scale (VAS) score was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of intravenous regional anesthesia
  Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and VAS score was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the OR and the performance of Intra-Venous regional Anesthesia (IVRA)
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 46 | 47
score on a scale | 1.22 (1.12) | 1.02 (1.24)

2. Secondary Outcome: Degree of Satisfaction
Description: To perceive any disparity in patient's satisfaction degree measured through final questionnaire. A satisfaction questionnaire with evaluation from 0 (min) to 10 (max) regarding this topics. Higher values represent the better outcome, lower values represent the worse outcome.
Time Frame: 3 hours
Population: Control group underwent a surgical pre-operative examination, during which they received detailed information about surgical procedure but not regarding anesthetic technique. Video group patients received the same preoperative preparation procedur, and also watched a video group patients showed a 6-minute educational information video about IVRA.
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 46 | 47
units on a scale (0-10)
  General environment | 9.38 (1.01) | 9.5 (0.83)
  Equipments | 9.5 (0.83) | 9.5 (1.02)
  Organization of departments | 9.61 (0.75) | 9.51 (0.83)
  Waiting list | 8.56 (2.15) | 8.84 (1.81)
  Pharmacy Service | 9.42 (1.13) | 9.55 (1.09)
  Nursing professionals | 9.68 (0.6) | 9.68 (1.04)
  Medical professionalism | 9.9 (0.29) | 9.73 (1.06)
  Informations | 9.86 (0.34) | 9.72 (0.79)
  Time dedicated to patient | 9.76 (0.47) | 9.5 (1.13)

3. Secondary Outcome: Vital Parameters 1: Arterial Blood Pressure
Description: To see any variance in vital parameters that are usually affected by anxiety, like arterial blood pressure [mmHg] in all patients.
Time Frame: 2 hours
Population: Systolic arterial pressure measured on admission in the day-hospital clinic.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 46 | 47
mmHg
  Systolic Arterial Pressure | 139.36 (22.08) | 129.17 (17.8)
  Diastolic Arterial Pressure | 81.69 (10.9) | 78.43 (10.12)

4. Secondary Outcome: Vital Parameters 2: Respiratory Rate
Description: To see any variance in vital parameters that are usually affected by anxiety like respiratory rate [breath per minute] in all patients.
Time Frame: 2 hours
Population: Respiratory rate at anesthesia
Measure: Mean (Standard Deviation); unit: breath per minute
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 46 | 47
breath per minute | 14.71 (3.07) | 13.86 (1.48)

5. Secondary Outcome: Vital Parameters 3: Heart Rate
Description: To see any variance in vital parameters that are usually affected by anxiety like heart rate [beat per minute] in all patients.
Time Frame: 2 hours
Population: Cardiac rate at anesthesia
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 46 | 47
bpm | 75.45 (13.08) | 71.76 (10.23)

6. Secondary Outcome: First Subgroups Analyze: Anxious Patients
Description: A subgroup analysis was performed applied to specific subgroups, like anxious patients.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and Visual Analog Pain Scale (VAS) was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the operating room and the performance of intravenous regional anesthesia
  Video Group: Patients in the film group watched the film using a laptop computer equipped with headphones, and VAS score was repeated after the movie. Video was recorded by the Anaesthesiology department team, in order to explain and show in a detailed way on a model, the sequence of events, which occurs between the arrival of patients in the OR and the performance of Intra-Venous Regional Anesthesia (IVRA)
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 15 | 13
mmHg
  Systolic arterial Pressure | 135 (33.04) | 138 (21.2)
  Diastolic Arterial Pressure | 83 (5.6) | 79 (11.13)

7. Secondary Outcome: Second Subgroups Analyze: Higher Anxiety Score
Description: A subgroup analysis was performed applied to specific subgroups, like patients with higher anxiety assessment result, identified to have 3 or more on the 5 point on Visual Analog Scale - Adapted (VAS-A) score (ranging from 1 - no anxious - to 5 - totally anxious).
Time Frame: 2 hours
Population: This analysis is made to see if video is ineffective in reducing anxiety level
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 16 | 10
mmHg
  Systolic Arterial Pressure | 129.36 (34.73) | 127.11 (10.74)
  Diastolic Arterial Pressure | 78.21 (13.9) | 72.7 (7.54)

8. Secondary Outcome: Third Subgroup Analyze: First Experience With Surgery.
Description: A subgroup analysis was performed applied to specific subgroups, like patients at their first experience with surgery, identified by specific questionnaire.
Time Frame: 2 hours
Population: A third subgroup analysis took into account patients for whom the operation was their first surgical experience.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Video Group | Control Group
Number analyzed (Participants) | 23 | 19
mmHg
  Systolic Arterial Pressure | 132.65 (32.56) | 129.82 (15.28)
  Diastolic Arterial Pressure | 80.8 (9.77) | 74.7 (11.1)

ADVERSE EVENTS:
Time Frame: 2 hours after surgical intervention
Description: The authors did not foresee the appearance of side effects after viewing the video.
Arm/Group | Video Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

LIMITATIONS AND CAVEATS:
* Authors adopted the VAS score.
* Type of surgery has been shown to influence anxiety levels.
* The study was not adequately powered to assess statistical significance of these secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT03581097/Prot_SAP_000.pdf